CLINICAL TRIAL: NCT02626117
Title: Laser De-epithelialization for Epithelial Exclusion in Root Coverage Procedure: a Clinical Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_36651
Record Dates: First submitted 2015-12-01; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAF+ SCTG+ laser depithelialisation (Active Comparator): CAF + SCTG and Diode (GaAlAs) laser with a wavelength of 820 nm and a power of 1.5 watt in a continuous mode was applied to remove the sulcular epithelium.
  Interventions: Device: LASER deepithelialization
- CAF+SCTG+ sham laser depithelialisation (Sham Comparator): CAF+ SCTG+ sham LASER deepithelialisation was applied to remove the sulcular epithelium.
  Interventions: Device: Sham LASER deepithelialization

INTERVENTIONS:
Device: LASER deepithelialization — the selected participants were assigned in test and control. Under LA full thickness flap was reflected until the mucogingival junction and recipient area was prepared. The connective tissue graft harvested from palate was placed on the root surface and secured with 5-0 absorbable sutures. Diode (GaAlAs) laser with a wavelength of 820 nm and a power of 1.5 watt in a continuous mode was applied to remove the sulcular epithelium. The connective tissue graft was placed on the root surface at the level of the CEJ and then secured with 5-0 absorbable sutures in both test and control sites using sling suture..
  Arms: CAF+ SCTG+ laser depithelialisation
Device: Sham LASER deepithelialization — the selected participants were assigned in test and control. Under LA full thickness flap was reflected until the mucogingival junction and recipient area was prepared. The connective tissue graft harvested from palate was placed on the root surface and secured with 5-0 absorbable sutures. sham LASER deepithelialisation was applied to the sulcular epithelium. The connective tissue graft was placed on the root surface at the level of the CEJ and then secured with 5-0 absorbable sutures in both test and control sites using sling suture..
  Arms: CAF+SCTG+ sham laser depithelialisation

SUMMARY:
The concept of laser deepithelialization to retard epithelial migration has enabled new attachment formation in periodontal pockets. Based on this hypothesis, that laser deepithelialization during root coverage procedures will enhance clinical outcome, a split mouth randomized controlled clinical trial was planned to compare the clinical outcome of Coronally advanced flap (CAF) + subepithelial connective tissue graft (SCTG) alone and in combination with laser de-epithelialization in the treatment of gingival recession.

DETAILED DESCRIPTION:
Successful treatment of recession defects to obtain new attachment and prevent repair by long junctional epithelium continues to present a serious therapeutic challenge. The concept of laser deepithelialization to retard epithelial migration has enabled new attachment formation in periodontal pockets. Based on this hypothesis, that laser deepithelialization during root coverage procedures will enhance clinical outcome, a split mouth randomized controlled clinical trial was planned to compare the clinical outcome of Coronally advanced flap (CAF) + subepithelial connective tissue graft (SCTG) alone and in combination with laser de-epithelialization in the treatment of gingival recession.

METHOD:

In a split-mouth study, 20 patients presenting at least one pair of bilaterally symmetrical Miller's Class I and Class II buccal gingival recessions will be selected. Control site will receive coronally advanced flap with connective tissue graft and test site will receive laser deepithelialization as an adjunct to coronally advanced flap with connective tissue graft. Gingival recession depth (GRD), Gingival recession width (GRW), Probing depth (PD), Clinical attachment level (CAL), Keratinized tissue width (KTW), Plaque index (PI), Gingival index (GI), Gingival bleeding index (GBI) will be measured at baseline, 6 weeks, 3 months and 6 months after treatment. The root coverage outcomes were also assessed by photogrammetric analysis.

ELIGIBILITY:
Inclusion Criteria:• Miller's Class I and II recession defects involving maxillary or mandibular canines or premolars.

* Similar bilateral recession defects.
* Systemically healthy patients.
* Patients willing to participate in study.
* Age group of 21-57 years.
* Patients with esthetic concerns.

Exclusion Criteria:

* Pregnant and lactating woman
* Patients who have undergone any type of regenerative periodontal therapy six months prior to the initial examination.
* Patients with history of smoking.
* Teeth with hopeless prognosis.
* Root surface restoration.

Ages: 21 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of root coverage (PRC) | 6 months
Complete root coverage | 6 months

SECONDARY OUTCOMES:
Reductions in recession depth (Rec Red) | 6 months
Gingival recession width (GRW) | 6 months
Probing depth (PD) | 6 months
Clinical attachment level (CAL) | 6 months
Keratinized tissue width (KTW) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joann Pauline George, MDS, Study Director — krishnadevaraya college of dental sciences
Locations (1):
- Dr Joann Pauline George, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nevins ML, Camelo M, Schupbach P, Kim SW, Kim DM, Nevins M. Human clinical and histologic evaluation of laser-assisted new attachment procedure. Int J Periodontics Restorative Dent. 2012 Oct;32(5):497-507. PMID 22754897
- See also: reference article — http://www.ncbi.nlm.nih.gov/pubmed